CLINICAL TRIAL: NCT05346341
Title: Evaluation of the Effect of Minimally Invasive Procedures Used in Management of Salivary Ductal Pathologies on Patients' Symptomatology and Gland Function - A Clinical Trial
Brief Title: Evaluation of the Effect of Minimally Invasive Procedures Used in Management of Salivary Ductal Pathologies on Patients' Symptomatology and Gland Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aya Sakr (Other)
Responsible Party: Sponsor-Investigator, Aya Sakr, Assistant Lecturer of Oral and Maxillofacial Surgery, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00010556 - 0008839
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Salivary Gland Stone; Salivary Gland Diseases
MeSH Terms: conditions — Salivary Gland Calculi; Salivary Gland Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally invasive techniques (Experimental)
  Interventions: Procedure: Minimally invasive techniques

INTERVENTIONS:
Procedure: Minimally invasive techniques — All patient will be treated under general anaesthesia An appropriate gland-preserving minimally-invasive surgical procedure will be performed for all patients according to the nature and extent of the disease for either submandibular or parotid ducts.
  Minimally invasive techniques for ductal salivary gland pathologies include:
  1. Sialolithotomy through a simple cutdown
  2. Sialendoscopy
  3. Transoral microscopic-assisted sialolithotomy.

SUMMARY:
Aim of the current study was to evaluate the minimally invasive techniques in the management of salivary gland ductal pathologies

ELIGIBILITY:
Inclusion Criteria:

* All patients manifesting with either submandibular or parotid salivary gland ductal pathologies including:
* Sialolithiasis (salivary stones).
* Salivary ductal stenosis or stricture.
* Children with juvenile recurrent parotitis.
* Sjogren's syndrome.
* Radio-iodine induced sialadenitis.

Exclusion Criteria:

* Patients who are unfit for surgery.
* Patients with previous submandibular or parotid surgical resection.
* Patients with salivary tumors either benign or malignant.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Subjective salivary gland performance | up to 12 months
  This was done using a questionnaire to measure salivary score (this questionnaire is formulated by the multidisciplinary salivary gland society "MSGS"). The questionnaire consists of 20 questions divided in two groups: 13 regarding xerostomia and 7 regarding sialadenitis. Each question is scored from 0 to 10 and the total score could vary from 0 to 200 points.
Objective salivary gland performance (salivary flow measurement) | up to 12 months
  We have chosen 6 minutes as our standard time to collect saliva and we have chosen on purpose to collect saliva separately from the two parotids and jointly from the submandibular gland. A 5cmx5cm gaze is applied on the papilla of each Stenson duct and a third one is placed under the tongue. All these tampons are weighted separately after 6 minutes and the results collected.

CONTACTS AND LOCATIONS:
Overall Officials: Aya Sakr, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt